CLINICAL TRIAL: NCT02761031
Title: Perioperative Heart Rate Variability Analysis in Realtime: Detection of Cardiovascular and Autonomic Dysfunction
Brief Title: Perioperative Heart Rate Variability Analysis in Realtime
Acronym: PHERVR
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Vienna University of Technology (Other)
Responsible Party: Principal Investigator, Adam Joel Bukaty, Dr. Adam Joel Bukaty, Medical University of Vienna
Other Study IDs: 2095/2015
Record Dates: First submitted 2016-05-02; First posted 2016-05-04 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Individuality; Perioperative/Postoperative Complications; Heart Rate and Rhythm Disorders; Surgical Complications From General Anesthesia
Keywords: Heart rate variability; Electrocardiography; Observational study; Non-interventional study; Risk assessment; Perioperative
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
This study will record patient electrocardiograms - as well as various other body signals (e.g., blood pressure, pulse wave, peripheral hemoglobin oxygen saturation) - as monitored routinely both during and immediately subsequent to surgical operations performed under general anesthesia. Through retrospective analysis of patients' heart rate variability (HRV), in concert with the other abovementioned parameters, the investigators seek to forward the development of novel mathematical models and tools for on-line detection of cardiovascular and autonomic dysfunction in the perioperative setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing non-cardiac surgery under general anesthesia
* Patients aged 18-80 years
* Patients who are capable of giving informed consent

Exclusion Criteria:

* Patients <18 or >80 years of age
* Patients with an active cardiac pace maker
* Patients with an absent sinus rhythm in ECG
* Patients presenting with a preexisting arrhythmia
* Patients requiring postoperative ICU therapy
* Patients with pheochromocytoma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients between the ages of 18 and 80 who are undergoing non-cardiac surgery under general anesthesia at Vienna General Hospital may participate.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2016-04; Primary Completion 2018-05 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | During and immediately subsequent to surgery performed under general anesthesia
  The analysis of heart rate variability (HRV) has been used to assess autonomic nervous system responses to therapeutic interventions, and to quantify risk in a wide variety of both cardiac and non-cardiac disorders when combined with other diagnostic tests - though HRV analysis has seen its greatest cardiologic use in post-myocardial infarction risk stratification and in assessing risk for arrhythmic events. HRV analysis has become widespread and relatively simple to perform - however, until now, these analyses have not been performed in detail in the perioperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Adam J Bukaty, MD, Principal Investigator — Medical University of Vienna; Ulrich Klein, MD, PD, Study Director — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria